CLINICAL TRIAL: NCT03663972
Title: Age-related Correlates of Treatment Efficacy and Efficiency for Late-acquired Sounds
Brief Title: Age-related Correlates of Treatment for Late-acquired Sounds
Acronym: ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Breanna Irene Krueger, Assistant Professor, University of Wyoming
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180510BK01978
Record Dates: First submitted 2018-08-31; First posted 2018-09-10 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Speech Sound Disorder; Phonology Disorder; Phonology Impairment; Phonological Disorder; Articulation Disorders in Children; Developmental Phonological Disorder; Speech Disorders; Speech Delay; Articulation Disorders, Developmental
Keywords: treatment; efficacy; efficiency; late-acquired sounds
MeSH Terms: conditions — Speech Sound Disorder; Articulation Disorders; Speech Disorders; Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Young children (age 4-5) and Old children (age 7-8) will be enrolled in either a Motoric behavioral treatment arm or phonological treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motoric Arm (Active Comparator): Children will participate in an intervention based on traditional articulation approaches to speech therapy.
  Interventions: Behavioral: articulation therapy
- Phonologic Arm (Active Comparator): Children will receive intervention that targets the conceptual representation of sounds.
  Interventions: Behavioral: phonologic treatment

INTERVENTIONS:
Behavioral: articulation therapy — children receive instruction in producing new sounds at the isolation, syllable and word level.
  Arms: Motoric Arm
Behavioral: phonologic treatment — children receive instruction in producing new sounds at the word level
  Arms: Phonologic Arm

SUMMARY:
Late-acquired sounds, such as /r/ are difficult to learn and many children experience persistent errors on these sounds. The purpose of the present study is to determine whether treating these sounds earlier in the child's life may result in better outcomes.

DETAILED DESCRIPTION:
Late-acquired sounds, such as /r/ are difficult to learn and many children experience persistent errors on these sounds. However, these sounds are often treated later in a child's life because they are not expected to be fully acquired until quite late--age 7-8 for some sounds. This practice places treatment in a time of the child's development in which they struggle to learn new sounds.The purpose of the present study is to determine whether treating these sounds earlier in the child's life may result in better outcomes, and to examine treatment efficacy and efficiency for two methods of treatment.

ELIGIBILITY:
Inclusionary Criteria:

* Normal Hearing
* Typical Receptive Language
* Speech Sound Disorder
* No motor speech impairment
* Typical non-verbal intelligence
* Produces at least one late-acquired sound with <7% accuracy
* Monolingual English-speaking
* Typical in terms of motoric and neurological development

Exclusionary Criteria:

* Neurological disorder
* Hearing loss
* Nonverbal IQ < 16th percentile

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Treatment Efficacy: Number of correct productions of treated speech sounds in treatment words | baseline until accuracy criterion is met; up to 18 weeks after final baseline session
  Accurate Production of treatment sound at baseline and at posttest
Treatment Efficiency: Number of sessions required to meet accuracy criteria | baseline until accuracy criterion is met; up to 18 weeks after final baseline session
  Number of treatment sessions required to meet accuracy criteria (90% accuracy across three consecutive sessions or a maximum of 35 treatment sessions)
Session Length: Mean duration of sessions in minutes | First treatment session until final treatment session. Final treatment session occurs when accuracy of treatment sound is met (90% accuracy across three consecutive sessions or a maximum of 35 treatment sessions)
  Start and end time of session is recorded on scoresheet, then number of minutes for each session for each participant is found and the mean across all sessions is calculated.

SECONDARY OUTCOMES:
Accuracy of production of untreated sounds measured on pretest and posttest probes | baseline and at posttest up to 18 weeks after final baseline session
  Some children may generalize their skills learned through treatment to sounds that were not treated in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Breanna I. Krueger, PhD, Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krueger BI, Storkel HL. The impact of age on the treatment of late-acquired sounds in children with speech sound disorders. Clin Linguist Phon. 2023 Sep 2;37(9):783-801. doi: 10.1080/02699206.2022.2093130. Epub 2022 Jul 8. PMID 35801558